CLINICAL TRIAL: NCT02850354
Title: Gas Exchange and Cardiovascular Kinetics of Regulation - Effects of Short Term Changes in Gravity
Acronym: GasEx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-A01258-41
Record Dates: First submitted 2016-04-21; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- anti-g maneuvers (Experimental): Before the first parabola, pulmonary function will be evaluated. Then during each weightlessness period the subject will be instructed either to stay at rest (control condition) or to perform anti-g maneuvers (4 times each): intermittent exhalation on exertion, lower limbs and abdomen muscular contraction, combined maneuver ('intermittent exhalation on exertion' + 'muscle contraction'). Before, the exhalation on exertion, the subject will close the airway after the mouthpiece by pushing on a button actuating a pneumatic valve.
  Each subject will be tested during 15 parabola where the anti-g maneuvers will be performed in randomized order. After the 15th parabola, pulmonary function will be again evaluated.
  Interventions: Other: anti-g maneuvers

INTERVENTIONS:
Other: anti-g maneuvers — investigate the effects of anti-g maneuvers on cardiovascular and respiratory tolerance to the push-pull-effect.

SUMMARY:
The regulation of the cardiovascular respiratory system after changing environmental conditions or changes in work rates are essential for cognitive as well as physical functioning. For decades, it is known that high level of headward acceleration (+Gz) impairs cardiovascular function that may cause loss of consciousness. Some "anti-g" maneuvers, such as muscle contraction of the lower extremities and buttocks or intermittent exhalation on exertion (i.e., exhalation against a closed airway) have been proved to increase tolerance to high +Gz.

Main objective of this experiment is to investigate the effects of anti-g maneuvers on cardiovascular and respiratory tolerance to the push-pull-effect.

Cardiovascular and respiratory functions will be evaluated with the following parameters: heart rate, stroke volume, cardiac output, blood pressure, oxygen uptake, carbon dioxide output, ventilation, breathing frequency, body core temperature.

Electromyography (EMG) will not be a judgment criteria but will be used to check the quality of 'muscle contraction' anti-g maneuver.

The main hypothesis is that anti-g maneuvers will increase cardiovascular and respiratory tolerance to the push-pull effect, especially when they are combined.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 20 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign.

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Treated or non-treated arterial hypertension
* Smoker
* Asthma
* Respiratory bacterial or viral infection
* Pregnant women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
heart rate | baseline
  during 15 parabola
cardiac output with ECG | baseline
  during 15 parabola
blood pressure | baseline
  during 15 parabola
oxygen uptake measured with a spirometer | baseline
  during 15 parabola
carbon dioxide output measured with a spirometer | baseline
  during 15 parabola
ventilation measured with a spirometer | baseline
  during 15 parabola
breathing frequency measured with a spirometer | baseline
  during 15 parabola
body core temperature measured with 2 temperature sensors - one on forehead and the other one chest | baseline
  during 15 parabola

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — UMR 1075 UFR de Médecine Caen
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No